CLINICAL TRIAL: NCT05016245
Title: A Multicentre, Prospective, Open-label, Randomized Controlled Trial on the Efficacy and Safety of TheraSphereTM (Yttrium-90 Glass Microspheres) Compared to Conventional Transarterial Chemoembolization (cTACE) in Chinese Patients With Inoperable Hepatocellular Carcinoma
Brief Title: MANDARIN (S6371)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S6371
Record Dates: First submitted 2021-08-09; First posted 2021-08-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Inoperable Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TheraSphere™ Yttrium-90 Glass Microspheres (Experimental)
  Interventions: Combination Product: TheraSphere™ Yttrium-90 Glass Microspheres
- conventional Transarterial Chemoembolization(cTACE) (Active Comparator)
  Interventions: Procedure: conventional Transarterial Chemoembolization(cTACE)

INTERVENTIONS:
Combination Product: TheraSphere™ Yttrium-90 Glass Microspheres — TheraSphere™ Yttrium-90 Glass Microspheres TheraSphere™ is steam sterilized and supplied in 6 standard dose sizes: 3 GBq, 5 GBq, 7 GBq, 10 GBq, 15 GBq, 20 GBq. Custom dose sizes are also available in 0.5 GBq increments between 3 and 20 GBq.
  TheraSphereTM is supplied with the following accessories:
  Administration Set Administration Accessory Kit
  Arms: TheraSphere™ Yttrium-90 Glass Microspheres
Procedure: conventional Transarterial Chemoembolization(cTACE) — conventional Transarterial Chemoembolization(cTACE) is comprised of an anti-neoplastic agent(s) (i.e. cisplatin), lipiodol and embolic agent(s). The choice of agent(s) to be used is per usual local site practice. Chemotherapy agents can be as a single agent or used in combination, as per local practice.
  Arms: conventional Transarterial Chemoembolization(cTACE)

SUMMARY:
To evaluate the efficacy and safety of TheraSphereTM yttrium [90Y] glass microsphere in the Chinese patients with inoperable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 and ≤80 age and provided study consent
* Patients diagnosed with HCC and clinically evaluated as inoperable (as per local practice) or who refuse operation (ablation, hepatectomy and liver transplantation)
* At least one well defined HCC tumor measurable by mRECIST in contrast-enhanced MRI
* China liver cancer staging (CNLC) stage Ib~IIb
* Child-Pugh ≤ B7
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Tumor burden ≤50% of the total liver volume

Exclusion Criteria:

* Presence of extra-hepatic metastases or additional malignancies aside from HCC
* Patients with hepatic artery malformation and unable to intubate hepatic artery
* Patients who are allergic to contrast agents or have renal insufficiency (Serum creatinine>2mg/ml or Creatinine clearance<30mL/min) and are not suitable for injection of contrast agents
* Severe pulmonary insufficiency (FEV1/FVC<50% or FEV1/predicting value<50% or MVV<50L/min)
* AST and ALT >5 times upper limit of normal
* Clinical manifestations of decompensated cirrhosis (Grade2/3 of ascites, gastrointestinal bleeding, hepatic encephalopathy, etc. according to EASL Clinical Practice Guidelines)
* HCC invading biliary tract or causing biliary obstruction
* uncorrectable coagulation dysfunction and severe hemogram abnormality [Prothrombin time (PT)>6 seconds above control or PT-International normalized ratio (INR)>2.5, WBC<3.0x109/L, PLT<50x109/L]
* Infiltrative HCC tumor type
* Bilobar HCC disease
* Any presence of portal vein or hepatic veins or artery invasion
* Occlusion of portal vein completely with less collateral vessels
* Transjugular intrahepatic portosystemic shunt (TIPS) or Hepatic arterioportal fistula
* Patients during pregnancy or lactation
* Prior interventional therapy via hepatic artery or radiotherapy treatment for HCC
* Tc-99m macroaggregated albumin (MAA) hepatic arterial perfusion scintigraphy shows any deposition to the gastrointestinal tract that may not be corrected by angiographic techniques
* Radiation pneumonitis has been seen in patients receiving doses to the lungs greater than 30 Gy in a single treatment or greater than 50Gy in multiple treatment
* The absorbed dose of lung may exceed 30Gy in preoperative evaluation
* Receive any investigational therapy or anti-tumor therapy within 30 days prior to study enrollment
* Any other reason in which the investigator believes that the patient is unsuitable to participate in this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Time to progression (TTP) | through study completion, an average of 18 months
  Time to progression (TTP) Definition of progression: Progressive Disease (PD) assessment occurs according to mRECIST occurs according to mRECIST
Safety assessed within 60 days post treatment using NCI-CTCAE v5.0 | within 60 days post treatment
  Safety assessed within 60 days post treatment using NCI-CTCAE v5.0

SECONDARY OUTCOMES:
Hepatic time to progression (hTTP) determined by localized mRECIST (within the treated area) | through study completion, an average of 18 months
Objective response rate (ORR) of the index lesion according to localized mRECIST (within the treatment area) | through study completion, an average of 18 months
Confirmed ORR according to mRECIST | through study completion, an average of 18 months
OS (Overall Survival) | through study completion, an average of 18 months
Safety assessed using NCI-CTCAE v 5.0 | through study completion, an average of 18 months
  Safety assess: to standardize reporting, the National Cancer Institute Common Terminology Criteria (NCI CTCAE), version 5, was used to grade AEs and SAEs. Grades 1, 2, 3, and 4 represented mild, moderate, severe, and life-threatening toxicity, respectively. Grade 5 represented toxicity resulting in death. Descriptive analyses were conducted to assess the safety in each grade and summarized as the number of events and rate per subject.
Procedure technical success | immediately after the procedure
  Procedure technical success is determined successfully if all three items are satisfied at the same time during the operation as follow:
  * Device connected successfully or not;
  * Microspheres or anti-neoplastic agent(s) (i.e. cisplatin), lipiodol and embolic agent(s). deliver to target area well, or not by device parts;
  * There was no unplanned release of radiation or leakage of neoplastic agent(s) (i.e. cisplatin), lipiodol and embolic agent(s), or not by device parts.

CONTACTS AND LOCATIONS:
Overall Officials: Gaojun TENG, Dr., Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No